CLINICAL TRIAL: NCT02449993
Title: Evaluation of the MammaTyper Kit, Ref 90020/90021 Performed on Clinical Material Obtained From Patients With Early Breast Cancer: Re-Examination of Tumor Material and Re-Evaluation of Patient Data From Patients Treated With Neo-adjuvant Therapy
Brief Title: Re-Examination of Tumor Material and Re-Evaluation of Patient Data From Patients Treated With Neo-adjuvant Therapy
Status: Completed | Type: Observational
Sponsor: BioNTech Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MammaTyper_1.neo-adjuvant st.
Record Dates: First submitted 2015-05-06; First posted 2015-05-21 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: diagnostic study; analysis of estrogen receptor; progesterone receptor; Human epidermal growth factor receptor 2; Ki-67
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MammaTyper™: MammaTyper™ will be used to assess tumor material of patients treated with neo-adjuvant therapy.
  Interventions: Device: MammaTyper™

INTERVENTIONS:
Device: MammaTyper™ — MammaTyper™ is an in vitro molecular diagnostic test for the quantitative detection of the biomarkers estrogen receptor (ESR1), progesterone receptor ( PgR), Human epidermal growth factor receptor 2 (HER2) and proliferation antigen Ki-67 on the basis of the values of the messenger ribonucleic acid (mRNA).

SUMMARY:
This is a prospective examination of ribonucleic acid (RNA) extracted from tumor material of breast cancer patients treated with a neo-adjuvant therapy. The RNA will be analysed for expression of estrogen receptor (ER 1), progesterone receptor (PgR), HER2 and Ki-67 with MammaTyper™.

According to the determined values for the individual parameters at least 4 subtypes can be distinguished to date

* Luminal A-type
* Luminal B-type
* HER2-type
* Triple-negative-type As non-clinical endpoint, the agreement of new subtyping with Immunohistochemical methods will be evaluated.

As clinical objective, the 5 year Distant metastasis free survival (DMFS) and Overall survival (OS) will be reevaluated according to the new subtyping.

DETAILED DESCRIPTION:
Tumor material collected from patients who received neoadjuvant therapy either with four cycles of doxorubicin 60 mg/m² plus pemetrexed 500 mg/m² on day 1 every 21 days followed by four cycles of docetaxel 100 mg/m² on day 1 every 21 days or four cycles of doxorubicin 60 mg/m² plus cyclophosphamide 600 mg/m² on day 1 every 21 days followed by four cycles of docetaxel 100 mg/m² on day 1 every 21 days will be re-analyzed with the MammaTyper Kit. The Kit is an in-vitro molecular diagnostic test for molecular subtyping of breast cancers into Luminal A & B, HER2 and Triple negative. It allows quantitative detection of the RNA expression status of the genes for estrogen receptor (ESR1), PgR, HER2 and Ki-67 on the basis of their mRNA present in the samples. This prospective diagnostic study will investigate the subtyping-results of the MammaTyper™ analysis and will compare them to the subtyping of the former immunohistochemical analysis performed. Based on the MammaTyper™-subtypes the efficiency of the therapy regimen and the outcome will be re-evaluated from the patient data.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70 years with histologically confirmed primary invasive breast cancer stages T2-T4/N0-N2/M0 with a tumor size of ≥ 2 cm as measured by ultrasound
* The patient provides a written informed consent for analysis of tumor material

Exclusion Criteria:

* Prior anticancer therapy with an anthracycline or other prior antitumor therapy for breast cancer
* Inflammatory or exulcerating breast cancer
* A second primary malignancy [except carcinoma in situ (CIS) of the cervix or adequately treated nonmelanoma skin cancer] unless diagnosed and treated ≥ 5 years ago with no evidence of recurrence
* Any serious concomitant systemic disorder

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See Eligibility Criteria
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Agreement of new subtyping assessed as rate of patients in MammaTyper-subtype groups compared to rate of patients in subtype groups according to immunohistochemical analysis according to St. Gallen Guideline 2013 | Baseline
  For each MammaTyper and immunohistochemical based subtype categorization, percent agreement, positive and negative percent agreement as well as kappa-statistics are calculated.

SECONDARY OUTCOMES:
Assess difference of 5 year OS of breast cancer subgroup Luminal A vs. combined subgroup (Luminal B (HER2 positive / HER2 negative), HER2 positive, triple negative), based on subtyping with MammaTyper™ | 5 years from the date of patient registration
  Assessed as rate of patients in subgroup Luminal A with 5 year OS vs. rate of patients in combined subgroups with 5 year OS based on MammaTyper subtyping
Estimation of difference in prediction of pathologic complete remission for MammaTyperTM Ki-67 vs. local Ki-67 visual scoring assessment for Luminal tumors, whereby a positive difference is expected | Baseline
  Assessed as rate of patients with complete response and Ki-67 determination according to MammaTyper and visual scoring assessment
ESR1 mRNA is predictive for 5 year OS with low expression of ESR1 mRNA being associated with adverse outcome (rate of patients with 5 year OS and high or low expression of ESR1 mRNA) | 5 years from the date of patient registration
  Assessed as rate of patients with 5 year OS and high or low expression of ESR1 mRNA